CLINICAL TRIAL: NCT04337736
Title: The Impact of Different Physical Exercise Protocols on Cardio-vascular Efficiency and Quality of Life in Breast Cancer Survivors
Brief Title: Effects of Physical Exercise on Cardio-vascular Efficiency and Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Researcher, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCSPHE001
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer Female
Keywords: Physical exercise; Adherence to physical exercise; Global longitudinal strain; Ventricular-arterial coupling; Arterial stiffness; Epicardial fat thickness; Intima-media thickness; Endocrine therapy
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training (Active Comparator): 12-weeks, 3-days-a week, supervised aerobic (Nordic walking or Walking) physical exercise (PhE) protocol; duration of each PhE session: 70 minutes; rate of perceived exertion (RPE): 10-11 (1st-4th week); 12-13 (5th-8th week); 13-14 (9th-12th week).
  Interventions: Other: Physical exercise
- Resistance training (Active Comparator): 12-weeks, 2.3-days-a week (total of 28 lessons), supervised resistance physical exercise (PhE) protocol; duration of each PhE session: 50 minutes.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise

SUMMARY:
To examine the effects of different physical exercise protocols (aerobic training and resistance training) on cardio-vascular efficiency and quality of life in a population of breast cancer survivors (BCS), not treated with chemotherapy.

DETAILED DESCRIPTION:
The present study enrolled a population of BCS women who underwent surgical treatment for breast cancer at the "Ospedale G. Bernabeo" of Ortona, Chieti, Italy. The participants were randomized to the following physical exercise protocols: aerobic training, walking or Nordic walking; resistance training.

All the participants have been examined utilizing transthoracic echocardiography, carotid ultrasound and photo-plethysmographic method for the analysis of arterial stiffness, before and after the physical exercise protocol (T0-T1). The two-dimensional speckle-tracking analysis was performed with an offline, dedicated software from the apical 4-chambers-view. Moreover, ventricular-arterial coupling, epicardial fat thickness and intima-media thickness were also analyzed.

Quality of life was assessed using SF-36 score at T0, T1 and at a mean follow-up of 34 months. Moreover, at follow-up, we evaluated spontaneous physical activity and cardiovascular quality of life using IPAQ and SAQ-7 scores.

ELIGIBILITY:
Inclusion Criteria:

* age < 65 years;
* history of breast cancer surgery in the previous 12 months;
* no history of chemotherapy;
* no ongoing radiotherapy;
* eventual hormonal therapy;
* cardiovascular and orthopedic eligibility.

Exclusion Criteria:

* adjuvant chemotherapy;
* any history of cardiovascular disease;
* abnormal exercise stress test at the screening;
* any systemic inflammatory disease or any orthopedic condition potentially limiting the physical training.

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Improvement of cardio-vascular efficiency | 12-weeks (from the beginning of physical exercise training)
  A composite of the improvement in the following parameters, from pre-treatment values: global longitudinal strain analysis, as assessed by speckle-traking echocardiography; ventricular-arterial coupling, as assessed by echocardiographic single beat method; arterial stiffness (pulse wave velocity, augmentation index), as assessed by photoplethysmographic method

SECONDARY OUTCOMES:
Epicardial fat thickness reduction | 12-weeks (from the beginning of physical exercise training)
  A reduction in epicardial fat thickness evaluated with echocardiographic method
Intima-media thickness reduction | 12-weeks (from the beginning of physical exercise training)
  A reduction in epicardial fat thickness evaluated with ultrasonographic method
Improvement of quality of life | 12-weeks (from the beginning of physical exercise training); a mean of 34 months from the enrollment
  An improvement of quality of life, from pre-treatment values, evaluated with the 36-Item Short Form Health Survey (minimum value: 0, associated with the worst quality of life; maximum value: 100, associated with the best quality of life)
Improvement of spontaneous physical activity | a mean of 34 months from the enrollment
  An improvement of spontaneous physical activity evaluated with International Physical Activity Questionnaire score (0-700 MET: low level of physical activity; 700-2519 MET: intermediate level of physical activity; > 2520 MET: high level of physical activity)
Improvement of cardiovascular quality of life | a mean of 34 months from the enrollment
  An improvement of quality of life evaluated with the Seattle Angina Questionnaire-7 score (minimum value: 0, associated with more symptoms and with the worst quality of life; maximum value: 100, associated with fewer symptoms and with the best quality of life) where higher scores indicate fewer symptoms and higher health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, MD, PhD, Principal Investigator — ITAB - Institute for Advanced Biomedical Technologies; Valentina Bucciarelli, MD, PhD, Principal Investigator — ITAB - Institute for Advanced Biomedical Technologies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zamorano JL, Lancellotti P, Rodriguez Munoz D, Aboyans V, Asteggiano R, Galderisi M, Habib G, Lenihan DJ, Lip GYH, Lyon AR, Lopez Fernandez T, Mohty D, Piepoli MF, Tamargo J, Torbicki A, Suter TM; ESC Scientific Document Group. 2016 ESC Position Paper on cancer treatments and cardiovascular toxicity developed under the auspices of the ESC Committee for Practice Guidelines: The Task Force for cancer treatments and cardiovascular toxicity of the European Society of Cardiology (ESC). Eur Heart J. 2016 Sep 21;37(36):2768-2801. doi: 10.1093/eurheartj/ehw211. Epub 2016 Aug 26. No abstract available. PMID 27567406
- [Background] Khosrow-Khavar F, Filion KB, Al-Qurashi S, Torabi N, Bouganim N, Suissa S, Azoulay L. Cardiotoxicity of aromatase inhibitors and tamoxifen in postmenopausal women with breast cancer: a systematic review and meta-analysis of randomized controlled trials. Ann Oncol. 2017 Mar 1;28(3):487-496. doi: 10.1093/annonc/mdw673. PMID 27998966
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Zhu G, Zhang X, Wang Y, Xiong H, Zhao Y, Sun F. Effects of exercise intervention in breast cancer survivors: a meta-analysis of 33 randomized controlled trails. Onco Targets Ther. 2016 Apr 13;9:2153-68. doi: 10.2147/OTT.S97864. eCollection 2016. PMID 27110131
- [Background] Scott JM, Nilsen TS, Gupta D, Jones LW. Exercise Therapy and Cardiovascular Toxicity in Cancer. Circulation. 2018 Mar 13;137(11):1176-1191. doi: 10.1161/CIRCULATIONAHA.117.024671. PMID 29530893